CLINICAL TRIAL: NCT07296354
Title: Randomized, Double-Blind Active-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of an ATP-Containing Parenteral Vitamin B Complex in Patients With Symptomatic Diabetic Polyneuropathy
Brief Title: Evaluation of an ATP-Containing Parenteral Vitamin B Complex in Patients With Symptomatic Diabetic Polyneuropathy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Egyptian International Pharmaceutical Industries Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABOVE; ABOVE-2501 (Other: Egyptian International Pharmaceutical Industries Co. (EIPICO))
Record Dates: First submitted 2025-11-25; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Adenosine Triphosphate; Vitamin B Complex

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epinosine - B Forte Lyophilized (Active Comparator): The investigational medicinal product is Epinosine B Forte, a parenteral formulation administered by intramuscular injection
  Interventions: Drug: adenosine triphosphate
- vitamin B complex only (Placebo Comparator): The active control is a vitamin B-complex injectable formulation that does not contain ATP; manufactured by the sponsor specifically for clinical trial use only
  Interventions: Drug: Vitamin B Complex

INTERVENTIONS:
Drug: adenosine triphosphate — Each lyophilized ampoule contains:
  Adenosine Triphosphate (ATP) - 10 mg Cocarboxylase (Vitamin B1 derivative) - 50 mg Nicotinamide (Vitamin B3) - 20 mg Vitamin B12 (Cyanocobalamin) - 500 mcg
  Arms: Epinosine - B Forte Lyophilized
Drug: Vitamin B Complex — Each ampoule contains:
  Cocarboxylase 50 mg Vitamin B12 500 mcg Nicotinamide 20 mg
  Arms: vitamin B complex only

SUMMARY:
Epinosine B Forte ampoule is an intramuscular injectable supplement containing adenosine triphosphate (ATP), Cocarboxylase (vitamin B1 derivative), vitamin B12, and nicotinamide (vitamin B3). It is used to support nerve function, treat B vitamin deficiencies, enhance cellular energy metabolism, and alleviate symptoms of fatigue, neuropathy, and general weakness. Commonly prescribed for conditions like peripheral neuritis and recovery from nerve-related disorders. Side effects are generally mild and may include local injection site reactions or allergic responses. Clinical evaluation of this investigational product may provide valuable evidence for its efficacy in treating diabetic neuropathy where impaired energy metabolism and micronutrient deficits often coexist. Establishing the efficacy and safety of Epinosine B Forte through a structured clinical trial is therefore essential. Demonstrating clinical benefit would not only inform and optimize current treatment protocols for DPN but also support the potential for broader clinical application which includes routine use in diabetic care, integration into treatment guidelines, and possible extension to other neuropathic conditions where metabolic support may play a therapeutic role

DETAILED DESCRIPTION:
To evaluate the effectiveness of the IMP (Epinosine - B Forte Lyophilized Ampoules) compared to an active control (vitamin B complex only) in improving neuropathic symptoms in patients with symptomatic diabetic polyneuropathy based on a validated neurological symptom scoring system.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age at time of consent
2. Able to provide informed consent for study participation.
3. Diagnosed with either Type 1 or Type 2 diabetes mellitus, with glycated hemoglobin (HbA1c) ≤ 10%
4. Diagnosed with diabetic polyneuropathy, defined as a Diabetic Neuropathy Symptom (DNS) score ≥ 2, with symptom duration of at least 3 months prior to providing informed consent.
5. Willingness to comply with study procedures and attend scheduled study visits
6. Patients should be on a stable antidiabetic medication regimen for 30 days prior to randomization.

Exclusion Criteria: -

1. Non-diabetic causes of neuropathy, e.g., alcohol abuse, vitamin B12 deficiency, renal failure, or chemotherapy-induced neuropathy other diseases that causes presence of any severe pain associated with conditions other than DPN that may confuse or confound the assessment of neuropathic pain.
2. Current or recent (within 30 days from screening visit) use of Neuropathic pain treatments, including:

   2.1 Gabapentinoids (gabapentin, pregabalin),

   2.2Serotonin-norepinephrine reuptake inhibitors (duloxetine, venlafaxine, desvenlafaxine)

   2.3 Tricyclic antidepressants (e.g., amitriptyline) 2.4 Topical capsaicin preparations 2.5 Carbamazepine, 2.6 Oxcarbazepine, 2.7 Lamotrigine 2.8 topiramate 2.9 other agents for neuropathic pain , Sedatives and anxiolytics (Benzodiazepines, Z-drugs (e.g., zolpidem), Barbiturates, Other B-complex or ATP-containing injectable supplements 2.10 Multivitamins or nutritional supplements 2.11 Pentoxifylline or Naftidrofuryl oxalate, Alpha-lipoic acid or other drug classes indicated for treatment of neuropathic pain.
3. Severe comorbidities (e.g., malignancy, liver failure, end-stage renal disease, decompensated heart failure)
4. Pregnancy or breastfeeding
5. Female patients of childbearing potential not using effective contraception (e.g., oral contraceptives, DMPA, IUD, double barrier, sterilization, or confirmed postmenopausal status)
6. Known hypersensitivity to any component of the investigational product
7. Participation in another clinical trial within the past 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2028-02-10 (Estimated); Study Completion 2029-01-10 (Estimated)

PRIMARY OUTCOMES:
To compare the mean change in Diabetic Neuropathy symptoms Score (DNS) from baseline to week 12 between the two study arms | 12 weeks
  A simplified scoring system, the diabetic neuropathy symptom score (DNS) frequently used in clinical trials and medical practice , assessing pain, numbness, tingling and ataxia. The maximum score of DNS is four points, one point or more indicates neurological abnormalities . It was reported to be validated, fast and easy to perform, with a high predictive value when screening for diabetic polyneuropathy . DNS was found to be the most and modified NDS had equal specificity (100%). DNS had a better diagnostic efficacy (70 %) ]sensitive test (65.4%)

SECONDARY OUTCOMES:
Neuropathy- and foot ulcer-specific quality of life (Neuro-QoL) | 12 weeks
  Neuro-QoL (Quality of Life in Neurological Disorders) is a validated patient-reported outcome measurement system developed to assess the physical, mental, and social health-related quality of life (HRQoL) in individuals living with neurological conditions. It is applicable across various disorders, including diabetic polyneuropathy.
  The version used in this study consists of 35 items, grouped into the following components:
  * 27 items covering six life domains: o Pain (7 items)
    * Loss or reduction of sensitivity (3 items)
    * Diffuse sensory-motor symptoms (3 items)
    * Limitations in daily activities (3 items)
    * Interpersonal problems (4 items)
    * Emotional distress (7 items)
  * 6 global items, one appended to each domain (labeled A-F), assessing the overall perceived impact of that domain on HRQoL.
  * 2 final items: o One assessing the overall impact of foot problems on HRQoL.
    * One providing a general global rating of the participant's HRQoL.
Vibration perception threshold | 12weeks
  The VPT will be tested on the pulp of the large toe of either right or left foot. Average of three measurements will be taken to calculate the VPT value of the given patient. Values will be recorded in the CRF. The VPT values will be graded as 'normal' (<15v), 'mild' (15-20v), 'moderate' (20-25v) and >25 as 'severe' neuropathy ( Martin, C.L., et al.,, 2010).

IPD SHARING:
Plan to Share IPD: No